CLINICAL TRIAL: NCT00669864
Title: Effect of Biphasic Insulin Aspart 30 Combined With Metformin on Blood Glucose Control in Subjects With Type 2 Diabetes Inadequately Controlled With Basal Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1960
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp 30-30 (Experimental): Individual adjusted dose of biphasic insulin aspart 30 administered before breakfast and dinner in combination with metformin 1000-2000mg, up to three times daily
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Subcutaneous (under the skin) injection, twice daily
  Other Names: NovoMix® 30
Drug: metformin — Tablets, 1000 - 2000 mg daily

SUMMARY:
This trial is conducted in Asia. This single arm trial aims to evaluate the blood glucose control with twice daily biphasic insulin aspart 30 in combination with metformin in Chinese subjects with type 2 diabetes inadequately controlled with once or twice daily basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with basal insulin once or twice daily with or without oral anti-diabetic drugs (OADs) for at least 3 months
* HbA1c (glycosylated haemoglobin A1c) within the range of 7.5% to10.0% ( both inclusive)
* BMI (Body Mass Index) maximum 40 kg/m2

Exclusion Criteria:

* Metformin contraindications according to local practice
* Systemically treated with TZDs (thiazolidinediones) for more than one month within 6 months prior to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 sites in China
Pre-assignment Details: Eligible subjects, treated with basal insulin, stopped their oral anti-diabetic drug treatment and started a run-in period of forced metformin titration. Subjects on current metformin therapy could go through a modified titration. Doses were up-titrated weekly until either the max tolerated dose of at least 1500mg/day or a max dose of 2000mg/day.
Period: Overall Study
Arm/Group | BIAsp 30-30
Started | 293
Completed | 284
Not Completed | 9
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 293
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Previous treatment [Number; unit: Participants]
  Basal insulin analogue | 122
  Basal human insulin | 169
  Animal insulin | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI (Body Mass Index) measured at baseline (week 0)
  kg/m^2 | 24.89 (3.28)
Duration of diabetes [Mean (Standard Deviation); unit: Years] — Number of years since diagnosis
  Years | 8.54 (5.49)
HbA1c [Mean (Standard Deviation); unit: percentage (%) of total haemoglobin] — HbA1c (Glycosylated Haemoglobin A1c) at baseline (week 0)
  percentage (%) of total haemoglobin | 8.16 (0.89)
Weight [Mean (Standard Deviation); unit: kg] — Weight measured at baseline (week 0)
  kg | 68.1 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin A1c)
Description: Change in Glycosylated Haemoglobin A1c (HbA1c) from baseline (week 0) to 16 weeks (end of treatment)
Time Frame: week 0, week 16
Population: Intention-to-Treat analysis set (ITT) is all subjects who entered the trial treatment period and exposed to at least one dose of trial product.
Measure: Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
percentage (%) of total haemoglobin | -1.303 (0.056)
Statistical Analysis 1: Comparison: BIAsp 30-30; The null hypothesis (H0): HbA1c after 16 weeks - HbA1c at baseline ≥ 0% against the alternative hypothesis (H1): HbA1c after 16 weeks - HbA1c at baseline < 0%. If H0 rejected at a significance level of 2.5%, declare a significant mean HbA1c decrease; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — A significant mean HbA1c decrease was to be declared if H0 is rejected at a significance level of 2.5%; Estimated mean = -1.303, 95% CI [-1.414 to -1.192], Standard Error of Mean 0.056

2. Secondary Outcome: Change in 8-point Plasma Glucose Profile
Description: Summary of change in 8-point plasma glucose profile by week and time. The 8 time points measured were: Before each meal (breakfast, lunch and dinner), at 2 hours after each meal (breakfast, lunch and dinner), at bedtime, and at 3 AM, measured over 16 weeks of treatment
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
mg/dL
  Before breakfast, N=282 | -1.95 (0.15)
  2 hours after breakfast, N=282 | -3.69 (0.25)
  Before lunch, N=279 | -2.60 (0.22)
  2 hours after lunch, N=282 | -2.67 (0.24)
  Before dinner, N=282 | -2.38 (0.22)
  2 hours after dinner, N=281 | -3.63 (0.27)
  Bedtime, N=279 | -3.10 (0.24)
  3 AM, N=279 | -2.23 (0.18)

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Less Than 7.0%
Description: Percentage of subjects achieving the treatment target of a glycosylated haemoglobin A1c (HbA1c) level below 7.0% after 16 weeks of treatment
Time Frame: week 16
Population: Intention-to-Treat analysis set (ITT) using LOCF (Last Observation Carried Forward) is all subjects who entered the trial treatment period and exposed to at least one dose of trial product.
Measure: Number; unit: percentage of participants
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
percentage of participants | 60.4

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Below or Equal to 6.5%
Description: Percentage of subjects achieving the treatment target of a glycosylated haemoglobin A1c (HbA1c) level below or equal to 6.5% after 16 weeks of treatment
Time Frame: week 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
percentage of participants | 38.9

5. Secondary Outcome: Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes experienced in the trial from week 0 (baseline) to week 16 (end of treatment). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no plasma glucose or blood glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: weeks 0-16
Population: Safety analysis set consists of all subjects who entered the trial treatment period and exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
episodes
  Major | 0
  Minor | 39
  Symptoms only | 203

6. Secondary Outcome: Hypoglycaemic Episodes, Diurnal/Nocturnal
Description: Total number of hypoglycaemic episodes experienced in the trial from week 0 (baseline) to week 16 (end of treatment) during the day (diurnal) and the night (nocturnal).
Time Frame: weeks 0-16
Population: as for outcome 5
Measure: Number; unit: episodes
Arm/Group | BIAsp 30-30
Number analyzed (Participants) | 293
episodes
  Diurnal | 188
  Nocturnal | 34
  Start time missing | 20

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time span of 16 weeks.
Description: Safety analysis set consists of all subjects who entered the trial treatment period and exposed to at least one dose of trial product.
Arm/Group | BIAsp 30-30
Serious Adverse Events (participants affected / at risk) | 0/293
Other Adverse Events (participants affected / at risk) | 80/293
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30-30 (N=293)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 4 (4)
Adverse drug reaction (General disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6)
Hypersensitivity (Immune system disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (21)
Otitis externa (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood triglycerides abnormal (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 2 (2)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Electrocardiogram ST-T segment abnormal (Investigations) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 2 (2)
Lipids abnormal (Investigations) | 3 (3)
Lipids increased (Investigations) | 1 (1)
Low density lipoprotein abnormal (Investigations) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 (14)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Vascular headache (Nervous system disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This single-armed trial does not permit a comprehensive comparison between BIAsp30 and basal insulin. Otherwise, this could have proffered greater clarity on the putative benefits that BIAsp30 brings to subjects with type 2 diabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.